CLINICAL TRIAL: NCT06021093
Title: HYPNotherapy for Improving Distress and Sleep in Adolescents and Young Adults With Cancer; a Feasibility Study (HYPNAYA Feasibility Study)
Brief Title: HYPNAYA Feasibility Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Jacqueline M. Tromp, Principal Investigator, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: NL83528.018.23
Record Dates: First submitted 2023-08-23; First posted 2023-09-01 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: AYA Cancer Patients
Keywords: Medical Hypnosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Medical Hypnosis: Study intervention: The hypnotherapy will include 2 individual hypnotherapy sessions plus daily listening to these recorded sessions and to (3 or 4) standardized hypnosis recordings. The individual sessions will be provided by CF and ET, both certified hypnotherapists and health care professionals (respectively nurse and physician). Preferably, these sessions take place during a planned admission for chemotherapy. If preferred by the patient, this can also take place at the hypnotherapist's office. If preferred by the patient, this can also take place at the venue of the hypnotherapist. A large part of the first session will be devoted to answering participants' questions and giving information about hypnosis, followed by exercises as an introduction to hypnosis. The goal of these exercises is to enable participants to increase their awareness and abilities in accessing mental imagery and hypnosis. At the end of the session, information will be provided about the home-based practice.

SUMMARY:
Adolescents and young adults (AYAs) with a cancer diagnosis experience high levels of stress during and after treatment. Hypnotherapy as supportive treatment throughout regular cancer care may reduce symptoms of distress, and improve sleep and health-related quality of life in AYAs with cancer. The objective of this pilot study is to demonstrate feasibility of hypnotherapy as supportive treatment.

DETAILED DESCRIPTION:
Study design: The HYPNAYA feasibility study is an interventional prospective single center cohort study with pre- and post-measurements. Patients will be consecutively recruited at the medical oncology department of the Amsterdam UMC. Participants will receive two hypnotherapy sessions including homebased exercises. At baseline, 8 and 12 weeks after the first hypnotherapy session, patients will be asked to fill in questionnaires.

Study population: consecutive AYAs (age 18-39) at the (outpatient) clinic undergoing systemic treatment or follow-up up to 6 months after finishing medical treatment. Patients that are actively treated by a psychiatrist, mentally incompetent (based on the opinion of the treating physician) or previously received hypnotherapy will be excluded.

Studie intervention: the hypnotherapy will include 2 individual hypnotherapy sessions plus daily listening to these recorded sessions and to (3 or 4) standardized hypnosis recordings. The individual sessions will be provided by CF and ET, both certified hypnotherapists and health care professionals (respectively nurse and physician). Preferably, these sessions take place during a planned admission for chemotherapy. If preferred by the patient, this can also take place at the hypnotherapist's office. If preferred by the patient, this can also take place at the venue of the hypnotherapist. A large part of the first session will be devoted to answering participants' questions and giving information about hypnosis, followed by exercises as an introduction to hypnosis. The goal of these exercises is to enable participants to increase their awareness and abilities in accessing mental imagery and hypnosis. At the end of the session, information will be provided about the home-based practice. This will consist of daily listening to prerecorded standardized hypnosis exercises for three months. These are standardized hypnosis excercises that will be specifically developed for this study and will be provided to all participants in the study. It will be explained that daily listening is essential to take full advantage of hypnosis without the help of a therapist. The second individual session will be scheduled 4-6 weeks later. During the second meeting, a new hypnosis exercise will be introduced and questions about the hypnotic exercises will be answered. Suggestions given during the hypnosis exercises will be focused on relaxation, improvement of sleep, more energy, ego-strengthening and improvement of feelings of anxiety and depression. It will again be explained that daily listening is essential to take full advantage of hypnosis without the help of a therapist.

ELIGIBILITY:
Inclusion criteria

* Consecutive AYA patients undergoing systemic treatment or follow-up up to 6 months after finishing medical treatment at the Amsterdam University Medical Centers in Amsterdam, will be invited to participate.
* The Dutch definition of AYA is patients aged 18-39 years at cancer diagnosis.
* All patients need to be fluent in Dutch
* Able to understand the informed consent form
* Willing to provide written informed consent.

Exclusion criteria

* Patients that are actively treated by a psychiatrist will not be able to participate in this study to prevent interference with ongoing psychiatric treatment.
* Patients that are mentally incompetent (based on the opinion of the treating physician) will be excluded.
* Patients that previously received hypnotherapy will also be excluded.

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Consecutive AYAs (age 18-39) at the (outpatient) clinic undergoing systemic treatment or follow-up up to 6 months after finishing medical treatment. Patients that are actively treated by a psychiatrist, mentally incompetent (based on the opinion of the treating physician) or previously received hypnotherapy will be excluded.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-07-17 (Actual); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility of hypnotherapy as supportive treatment for AYA patients | 8 weeks
  The primary outcome is feasibility of hypnotherapy as supportive treatment for AYA patients defined as the proportion of patients that complete the 8 weeks of treatment. Complete is defined as attending both individual hypnotherapy sessions.

SECONDARY OUTCOMES:
Feasibility of included questionnaires | 0, 8 and 12 weeks
  Feasibility of included questionnaires measured by the proportion of patients that complete all questionnaires pre-intervention (T0) and post-intervention (T3 and T4)
Feasibility of self-hypnosis | 8 and 12 weeks
  Feasibility of self-hypnosis measured by the proportion of patients that weekly perform self-hypnosis exercises and use recorded scripts for self-hypnosis measured using a structured exit interview on the experiences with medical hypnotherapy.
Patient-reported satisfaction of medical hypnosis | 8 and 12 weeks
  Patient-reported satisfaction of medical hypnosis measured using a structured exit interview on the experiences with medical hypnotherapy.
Reach of medical hypnosis | 1 year
  Reach measured as the number of participants and non-participants from the eligible patient population. Both numbers are retrieved from the central study database completed by the study coordinator.
Distress (i.e. anxiety) | 0, 8 and 12 weeks
  Distress (i.e. anxiety) measured using the Patient-Reported Outcomes Measurement Information System (PROMIS) Anxiety (8a) questionnaire (range 8 to 40, higher scores indicate higher level of anxiety).
Distress (i.e. depression) | 0, 8 and 12 weeks
  Distress (i.e. depression) measured using the Patient-Reported Outcomes Measurement Information System (PROMIS) Depression (8a) questionnaire (range 8 to 40, higher scores indicate higher level of depression).
Fear of cancer progression | 0, 8 and 12 weeks
  Fear of cancer progression as assessed using the Cancer Worry Scale (CWS) questionnaire (range 6 to 24, higher scores indicate high fear of cancer recurrence).
Quality of sleep | 0, 8 and 12 weeks
  Quality of sleep as assessed by the Pittsburgh Sleep Quality Index (PSQI) questionnaire (range 0 to 21), higher scores indicate worse sleep quality).
Health-related quality of life | 0, 8 and 12 weeks
  Health-related quality of life as assessed using the European Organization for Research and Treatment of Cancer Quality of Life Questionnaires Core-30 item (EORTC QLQ-C30, version 3.0) questionnaire (range 0 to 100, higher scores indicate better quality of life)
Change in distress (i.e. depression) | 0, 8 and 12 weeks
  Change in distress (i.e. depression) measured using the Patient-Reported Outcomes Measurement Information System (PROMIS) Depression (8a) questionnaire (range 8 to 40, higher scores indicate higher level of depression) pre-intervention (T0) and post-intervention (T3).
Change in distress (i.e. anxiety) | 0, 8 and 12 weeks
  Change in distress (i.e. anxiety) measured using the Patient-Reported Outcomes Measurement Information System (PROMIS) Anxiety (8a) questionnaire (range 8 to 40, higher scores indicate higher level of anxiety) pre-intervention (T0) and post-intervention (T3).
Change in fear of cancer progression | 0, 8 and 12 weeks
  Change in fear of cancer progression as assessed using the Cancer Worry Scale (CWS) questionnaire (range 6-24, higher score indicate high fear of cancer recurrence) pre-intervention (T0) and post-intervention (T3).
Change in quality of sleep | 0, 8 and 12 weeks
  Change in quality of sleep as assessed by the Pittsburgh Sleep Quality Index (PSQI) questionnaire (range 0 to 21, higher scores indicate worse sleep quality) pre-intervention (T0) and post-intervention (T3).
Change in health-related quality of life | 0, 8 and 12 weeks
  Change in health-related quality of life as assessed using the European Organization for Research and Treatment of Cancer Quality of Life Questionnaires Core-30 item (EORTC QLQ-C30, version 3.0) measured by comparing outcomes of questionnaires (range 0 to 100, higher scores indicate better quality of life) pre-intervention (T0) and post-intervention (T3).

CONTACTS AND LOCATIONS:
Locations (2):
- Netherlands (2):
  - Amsterdam UMC, location VUMC, Amsterdam, North Holland
  - Amsterdam UMC, location AMC, Amsterdam, North Holland

IPD SHARING:
Plan to Share IPD: Undecided
No specific plans but open to interested colleagues/persons

REFERENCES:
- See also: Related Info — https://hypnose4comfort.nl/
- See also: Related Info — https://skills4comfort.nl/